CLINICAL TRIAL: NCT01549249
Title: Evaluation of the Cone Outer Segment Tips Line After Epiretinal Membrane Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyorin University (Other)
Responsible Party: Principal Investigator, Makoto Inoue, Associate professor, Kyorin University
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: KyorinEye007
Record Dates: First submitted 2012-03-06; First posted 2012-03-09 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-11

CONDITIONS: Epiretinal Membrane
Keywords: cone outer segment tips line; inner segment/outer segment junction line; optical coherence tomography; epiretinal membrane
MeSH Terms: conditions — Epiretinal Membrane | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- vitrectomy (No Intervention)
  Interventions: Device: optical coherence tomography

INTERVENTIONS:
Device: optical coherence tomography — spectral-domain optical coherence tomography
  Other Names: vitreous surgery

SUMMARY:
The recovery of the cone outer segment tips (COST) line after epiretinal membrane (ERM) surgery using spectral-domain optical coherence tomography (SD-OCT) was assessed.

DETAILED DESCRIPTION:
Epiretinal membrane (ERM) may cause decreased central vision or metamorphopsia. Pars plana vitrectomy with membrane peeling has become the standard treatment for epiretinal membrane. However, visual recovery or symptomatic relief is not always satisfactory in all eyes despite successful membrane removal. Spectral domain optical coherence tomography (SD-OCT) is a non-invasive imaging device for various vitreoretinal diseases. Cone outer segment tips (COST) line is a line observed between IS/OS line and RPE in SD-OCT. The investigators examined the correlation of visual acuity and the recovery of photoreceptor layer after ERM surgery, taking COST line into account as a new parameter

ELIGIBILITY:
Inclusion Criteria:

* Patients who received epiretinal membrane surgery between June, 2008, and November, 2010, at Kyorin Eye Center.
* Only eyes with postoperative follow-up period more than 6 months were included.

Exclusion Criteria:

* Eyes with secondary epiretinal membrane (previous history of uveitis, intraocular surgery, pre-operatively noted retinal breaks, etc.) were excluded.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 333 (Actual)
Dates: Start 2008-06; Primary Completion 2010-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
best-corrected visual acuity | one year

SECONDARY OUTCOMES:
Integrity and defect length of the photoreceptor layer detected by spectral-domain optical coherence tomography | one year

CONTACTS AND LOCATIONS:
Overall Officials: Makoto Inoue, MD, Principal Investigator — Kyorin Eye Center
Locations (1):
- Kyorin Eye Center, Mitaka, Tokyo, Japan

REFERENCES:
- [Derived] Itoh Y, Inoue M, Rii T, Hirota K, Hirakata A. Correlation between foveal cone outer segment tips line and visual recovery after epiretinal membrane surgery. Invest Ophthalmol Vis Sci. 2013 Nov 5;54(12):7302-8. doi: 10.1167/iovs.13-12702. PMID 24106115